CLINICAL TRIAL: NCT05776680
Title: The Effects of Multi-Psycho-Oncology Care Courses Through Remote Psychological Support, Emotional Awareness Situation Videos and Empathic Concern Intervention on Physical and Psychological Status, Self-Efficacy and Empathy in Oncology Nurses
Brief Title: The Effects of Multi-Psycho-Oncology Care Courses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202112219RINB
Record Dates: First submitted 2022-11-03; First posted 2023-03-20 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Psychological; Oncology; Empathy
Keywords: cancer; Oncology nurse; Psychological support; Empathy; Training course
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological Support Course (Experimental): 60-minute once or twice a week for 6 months of Initial Remote Psychological Support Course .
  Interventions: Other: Psychological support
- Control group (No Intervention): Participants in control group will receive usual course.

INTERVENTIONS:
Other: Psychological support — 60-minute once or twice a week for 6 months of Initial Remote Psychological Support Course .
  Arms: Psychological Support Course

SUMMARY:
When the patient's mood has not yet reached a moderate to high severity level, psychological support is usually provided by the clinical nurses. However, the result of past research showed that the needs of patients and their caregivers were not satisfied with the psychological level. Scholars pointed out that it may be related to factors such as excessive clinical workload or insufficient psychological support and care capacity. In addition, under the influence of COVID-19 in the past two years, medical staff are facing more physical and mental pressure. Oncology nurses have a heavy workload and are affected by the COVID 19 epidemic, which reflects that nurses need psychological support. Therefore, this study intends to reduce stress through remote physical and mental support activities, and use the Internet to intervene in guided relaxation and meditation. Considering the scheduling of clinical nurses, a remote and unstructured course content that does not require continuity will be selected, and then advanced to provide the empathetic care skills of oncology nurses.

ELIGIBILITY:
Intervention group

* Inclusion Criteria:
* Over 20 years old (inclusive)
* Oncology nurses currently working in clinical practice
* Exclusion Criteria:
* Those who are unwilling or unable to participate in this course training for a full one- year period.
* Those who have registered for the advanced oncology nursing course organized by the Society in the current year.

Control group

* Inclusion Criteria:
* Over 20 years old (inclusive)
* Oncology nurses currently working in clinical practice
* Those who have registered for the advanced oncology nursing course organized by the Society in the current year
* Exclusion Criteria:
* Those who have participated in multiple oncology psychological care courses, those who are unwilling or unable to participate in the training of distance psychological support courses for a full one-year period.
* Those who participate in the advanced course of oncology nursing are unwilling or unable to participate in the data evaluation of the complete bi-annual time point.
* Those who have participated in this research project.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical and Psychological Symptoms Scale | 2 time points: Time 1 (before the psychological support course) ; Time 2 ( 6 months after the psychological support course)
  Oncology nurses' physical and psychological state were measured by physical and psychological state survey. It use Numerical Rating Scale(VRS) 0-10. It is a 11 Point Likert Scale (e. g. 0 is no pain; 10 is unbearable pain).

SECONDARY OUTCOMES:
Self efficacy scale (GSES) | 2 time points: Time 1 (before the psychological support course) ; Time 2 ( 6 months after the psychological support course)
  Oncology nurses' self-efficacy were measured by self efficacy scale. There are 10 questions about the level of confidence in these situations. It's a 4 point (1-4),higher the score means the more confident you have. There is also 11 point (0-10) scale that higher the score means the more confident you are in caring for patients.
Communication ability scale | 2 time points: Time 1 (before the psychological support course) ; Time 2 (6 months after the psychological support course)
  Oncology nurses' communication skills were measured by communication ability scale.It is a 5 Liker scale(1-5),higher scores represent better communication skills.
Efferson Empathy Scale | 2 time points: Time 1 (before the psychological support course) ; Time 2 ( 6 months after the psychological support course)
  Oncology nurses' empathy were measured by Efferson Empathy Scale. It is a 7 Liker scale(1-7),higher scores means someone have more empathy.
Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being （FACIT-Sp） | 2 time points: Time 1 (before the psychological support course) ; Time 2 ( 6 months after the psychological support course)
  Oncology nurses' spiritual well-being were measured by FACIT-Sp.It is a 5 Liker scale(0-4),higher scores represent better well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan